CLINICAL TRIAL: NCT03877900
Title: A Feasibility Study of Virtopsy With Tissue Sampling in Besancon University Hospital
Acronym: VIRTOPSY+
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/394
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Stillbirth and Fetal Death; Termination of Pregnancy; Neonatal Death
Keywords: post mortem Magnetic Resonance Imaging; stillbirth; fetal death; neonatal death; Minimally Invasive Autopsy; Tissue samplings
MeSH Terms: conditions — Stillbirth; Fetal Death; Perinatal Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to assess the feasibility of a new local post mortem procedure at Besançon University Hospital : Virtopsy+, magnetic resonance (MR) imaging with tissue sampling of the fetus and newborns.

DETAILED DESCRIPTION:
Minimally invasive autopsy is an alternative for conventional autopsy including post mortem magnetic resonance (MR) imaging and tissues samplings.

Because of the raise of parental refusal of autopsy, we intend to assess the local feasibility of a minimally invasive autopsy approach using post mortem MR imaging of fetuses and newborns in order to detect the major pathological abnormalities and/or to determinate the cause of death.

ELIGIBILITY:
Inclusion Criteria:

* stillbirth and fetal deaths over 21 weeks of gestation
* termination of pregnancy over 21 weeks of gestation
* neonatal death
* patient having read the letter of information and signed the consent.

Exclusion Criteria:

* legal incapacity
* limited ability to consent
* lack of parental consent

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * stillbirth and fetal deaths over 21 weeks of gestation
  * termination of pregnancy over 21 weeks of gestation
  * neonatal death
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Number of virtopsy made completely | month 12
  Number of virtopsy made completely (from death until clinical report).

CONTACTS AND LOCATIONS:
Overall Officials: Marion AUBER LENOIR, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addison S, Arthurs OJ, Thayyil S. Post-mortem MRI as an alternative to non-forensic autopsy in foetuses and children: from research into clinical practice. Br J Radiol. 2014 Apr;87(1036):20130621. doi: 10.1259/bjr.20130621. PMID 24288400
- [Background] Brookes JA, Hall-Craggs MA, Sams VR, Lees WR. Non-invasive perinatal necropsy by magnetic resonance imaging. Lancet. 1996 Oct 26;348(9035):1139-41. doi: 10.1016/S0140-6736(96)02287-8. PMID 8888168
- [Background] Breeze AC, Jessop FA, Set PA, Whitehead AL, Cross JJ, Lomas DJ, Hackett GA, Joubert I, Lees CC. Minimally-invasive fetal autopsy using magnetic resonance imaging and percutaneous organ biopsies: clinical value and comparison to conventional autopsy. Ultrasound Obstet Gynecol. 2011 Mar;37(3):317-23. doi: 10.1002/uog.8844. PMID 20878677
- [Background] Kang X, Cannie MM, Arthurs OJ, Segers V, Fourneau C, Bevilacqua E, Cos Sanchez T, Sebire NJ, Jani JC. Post-mortem whole-body magnetic resonance imaging of human fetuses: a comparison of 3-T vs. 1.5-T MR imaging with classical autopsy. Eur Radiol. 2017 Aug;27(8):3542-3553. doi: 10.1007/s00330-016-4725-4. Epub 2017 Jan 23. PMID 28116518
- [Background] Cannie M, Votino C, Moerman P, Vanheste R, Segers V, Van Berkel K, Hanssens M, Kang X, Cos T, Kir M, Balepa L, Divano L, Foulon W, De Mey J, Jani J. Acceptance, reliability and confidence of diagnosis of fetal and neonatal virtuopsy compared with conventional autopsy: a prospective study. Ultrasound Obstet Gynecol. 2012 Jun;39(6):659-65. doi: 10.1002/uog.10079. Epub 2012 May 22. PMID 21919100
- [Background] Griffiths PD, Paley MN, Whitby EH. Post-mortem MRI as an adjunct to fetal or neonatal autopsy. Lancet. 2005 Apr 2-8;365(9466):1271-3. doi: 10.1016/S0140-6736(05)74816-9. PMID 15811461
- [Background] Sebire NJ, Weber MA, Thayyil S, Mushtaq I, Taylor A, Chitty LS. Minimally invasive perinatal autopsies using magnetic resonance imaging and endoscopic postmortem examination ("keyhole autopsy"): feasibility and initial experience. J Matern Fetal Neonatal Med. 2012 May;25(5):513-8. doi: 10.3109/14767058.2011.601368. Epub 2011 Aug 10. PMID 21740313
- [Background] Woodward PJ, Sohaey R, Harris DP, Jackson GM, Klatt EC, Alexander AL, Kennedy A. Postmortem fetal MR imaging: comparison with findings at autopsy. AJR Am J Roentgenol. 1997 Jan;168(1):41-6. doi: 10.2214/ajr.168.1.8976917.
- [Background] Thayyil S, Sebire NJ, Chitty LS, Wade A, Olsen O, Gunny RS, Offiah A, Saunders DE, Owens CM, Chong WK, Robertson NJ, Taylor AM. Post mortem magnetic resonance imaging in the fetus, infant and child: a comparative study with conventional autopsy (MaRIAS Protocol). BMC Pediatr. 2011 Dec 22;11:120. doi: 10.1186/1471-2431-11-120. PMID 22192497
- [Background] D'Hondt A, Cassart M, De Maubeuge R, Soto Ares G, Rommens J, Avni EF. Postmortem fetal magnetic resonance imaging: where do we stand? Insights Imaging. 2018 Aug;9(4):591-598. doi: 10.1007/s13244-018-0627-0. Epub 2018 Jun 4. PMID 29869137